CLINICAL TRIAL: NCT03256721
Title: A Randomized, Parallel Control, Exploratory Trial to Compare Apatinib Plus Chemotherapy Drug Versus Chemotherapy Drug as Second-line Treatment in Subjects With Advanced or Metastatic of the Non-small Cell Lung Cancer (NSCLC)
Brief Title: Compare Apatinib Plus Chemotherapy Drug Versus Chemotherapy Drug as Second-line Treatment in NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the enrollment was slow and exceeded the expected enrollment time
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SECGOLC003
Record Dates: First submitted 2017-08-16; First posted 2017-08-22 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2018-08

CONDITIONS: Nonsmall Cell Lung Cancer
Keywords: apatinib docetaxel pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib; Docetaxel; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Group A: Apatinib 500mg QD PO d1-21 + Docetaxel (75mg/m2 IV d1)/Pemetrexed (500 mg/m2 IV d1), q21d
  Group B: Docetaxel (75mg/m2 IV d1)/Pemetrexed (500 mg/m2 IV d1), q21d
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib+docetaxel/pemetrexed (Experimental): Apatinib 500mg QD PO d1-21+docetaxel(75mg/m2 IV d1)/pemetrexed(500 mg/m2 IV d1),q21d
  Interventions: Drug: Apatinib/docetaxel/pemetrexed
- docetaxel/pemetrexed (Active Comparator): docetaxel(75mg/m2 IV d1)/pemetrexed(500 mg/m2 IV d1),q21d
  Interventions: Drug: docetaxel/pemetrexed

INTERVENTIONS:
Drug: Apatinib/docetaxel/pemetrexed — Participants are randomly assigned to treatment group or control group
  Arms: Apatinib+docetaxel/pemetrexed
Drug: docetaxel/pemetrexed — Participants are randomly assigned to treatment group or control group
  Arms: docetaxel/pemetrexed

SUMMARY:
Apatinib, a novel targeted inhibitor of VEGF receptor 2 (VEGFR2), shows significant antitumor activity in the patients with GC. The purpose of this study is to determine whether apatinib plus chemotherapy drug can improve progression free survival compared with chemotherapy drug in patients with metastatic the non-small cell lung cancer who failed one lines of chemotherapy.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in world wild, especially non-small cell lung cancer (NSCLC). Detection and early intervention are difficult because pathogenesis of NSCLC is not yet entirely clear.Most of them are advanced or metastatic patients, so approach 3/4 NSCLC undergo chemotherapy. Fewer treatment options exist on NSCLC whom is wild type of EGFR. The patient did not benefit from the existing treatment regimen after first-line treatment. There is currently no effective drug to treat this group of patients.

Apatinib, a novel targeted inhibitor of VEGF receptor 2 (VEGFR2), shows significant antitumor activity in the patients with GC. The purpose of this study is to determine whether apatinib plus chemotherapy drug can improve progression free survival compared with chemotherapy drug in patients with metastatic the non-small cell lung cancer who failed one lines of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age：18~75 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. Subjects with histologically or cytologically confirmed locally advanced or advanced NSCLC who have previously received no more than one lines treatment before participating；
4. Subjects with at least one measurable lesion as defined by RECIST (version 1.1),which is confirmed by computed tomography (CT) scan or MRI .
5. EGFRˉ,and ALK mutation in the negative or unknown；
6. Subjects without brain metastases or asymptomatic brain metastases, and not needing for dehydrating agents or corticosteroids to control intracranial symptoms;
7. Survival expectation≥ 3 months;
8. The main organ function is normal;
9. Females of childbearing potential must be a pregnancy test in 7 days before participating ( including serum or urine), and the results were negative.
10. Subjects provided written informed consent before participating,Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

1. Small Cell Lung Cancer;
2. Subjects with symptomatic brain metastases;
3. Survival expectation < 3 months;
4. Blood transfusion is required in the first dose of drug treatment within 14 days ;
5. The interval of subjects had received chemotherapy, biotherapy, radiotherapy or other anticancer therapies in the first dose of drug treatment within 21 days(excluding palliative radiotherapy);
6. The risk of active bleeding;
7. Subjects with uncontrolled blood pressure with medication (140/90 mmHg)
8. Laboratory values and organ functions ： （1）Hematologic insufficiency:

   1. Hemoglobin (Hb)<8.5 g/dL，
   2. Absolute neutrophil count (ANC)≤1.5×109/L，
   3. Platelet count (PLT)< 100×109/L； （2）Insufficient liver function:

   <!-- -->

   1. Bilirubin > 1.5×the upper limit of normal (ULN)
   2. Alanine aminotransferase (ALT), or Aspartate aminotransferase (AST) >3.0×(ULN), When liver metastases,Bilirubin > 1.5×ULN, ALT or AST >5.0×(ULN.
   3. serum creatinine ≤1.0×（ULN）, or creatinine clearance > 50 mL/min( calculated per the Cockcroft and Gault formula) (3) Subjects with positive for HBV surfaceantigen ( HBsAg)or anti-hcv (4)Subjects with Interstitial lung disease (5)Insufficient renal function: serum creatinine≥ 1.5×（ULN）, or creatinine clearance <60 mL/min
9. impairment of heart function: (1)Left ventricular ejection fraction (LVEF) <45% (LVEF evaluation is not required for subjects have no history of congestive heart failure), (2)Unstable angina, (3)Severe arrhythmia, (4)NYHA III or IVgrade of congestive heart failure, (5) Subjects with miocardial infarction within the last 12 months before entering the trial, (6)Pericardial effusion,
10. Subjects with liver fibrosis or hepatic cirrhosis
11. (1)Subjects with other active malignancy (except for definitively treated non melanoma skin cancer,carcinoma in-situ of the cervix,or other cancers that are treated with curative treatment and have no signs of recurrence for at least 5 years ) , (2)Subjects with dysphagia,malabsorption,chronic gastrointestinal diseases,or other medical history may hinder compliance and / or experimental drug absorption,
12. Subjects with major surgery in the first dose of drug treatment within 28 days,
13. Subjects with positive foknown human immunodeficiency virus。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  To compare progression-free survival (PFS) in subjects treated with apatinib plus chemotherapy drug versus chemotherapy drug as a second-line treatment in whom with advanced or metastatic non-small cell lung cancer (NSCLC)

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou general hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu Z, Cai X, Xu Z, He Z, Lai J, Wang W, Zhang J, Kong W, Huang X, Chen Y, Shi Y, Shi X, Zhao Z, Ni M, Lin X, Chen S, Wu X, Chen W, Song Z, Huang C. Apatinib plus Chemotherapy as a Second-Line Treatment in Unresectable Non-Small Cell Lung Carcinoma: A Randomized, Controlled, Multicenter Clinical Trial. Oncologist. 2020 Nov;25(11):e1640-e1649. doi: 10.1634/theoncologist.2020-0519. Epub 2020 Jul 25. PMID 32533785